CLINICAL TRIAL: NCT04707248
Title: Phase I, Two-Part, Multi-Center, First-in-Human Study of DS-6000a in Subjects With Advanced Renal Cell Carcinoma and Ovarian Tumors
Brief Title: A Study of DS-6000a in Subjects With Advanced Renal Cell Carcinoma and Ovarian Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS6000-A-U101
Record Dates: First submitted 2020-12-16; First posted 2021-01-13 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Carcinoma; Ovarian Tumor
Keywords: Renal Cell Carcinoma; Ovarian Tumor; Raludotatug deruxtecan (R-DXd; DS-6000a)
MeSH Terms: conditions — Carcinoma, Renal Cell; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Participants with ovarian cancer (OVC) or renal cell carcinoma (RCC) will receive an intravenous infusion of R-DXd (starting dose 1.6 mg/kg).
  Interventions: Drug: DS-6000a
- Dose Expansion: Cohort B-1 (Experimental): Participants with RCC will receive an intravenous infusion of R-DXd at the RDE. Enrollment has ended for this cohort.
  Interventions: Drug: DS-6000a
- Dose Expansion: Cohort B-2 (Experimental): Participants with OVC will receive an intravenous infusion of R-DXd at the RDE.
  Interventions: Drug: DS-6000a

INTERVENTIONS:
Drug: DS-6000a — Intravenous administration at doses starting at 1.6 mg/kg on Day 1 of Cycle 1
  Other Names: R-DXd
  Arms: Dose Escalation
Drug: DS-6000a — Intravenous administration at RDE on Day 1 of Cycle 1
  Other Names: R-DXd
  Arms: Dose Expansion: Cohort B-1; Dose Expansion: Cohort B-2

SUMMARY:
This clinical trial will evaluate raludotatug deruxtecan (R-DXd; DS-6000a) in participants with advanced renal cell carcinoma (RCC) and ovarian cancer (OVC). The main goals of this study will be to investigate the recommended dose of R-DXd that can be given safely to participants, assess the adverse events of R-DXd, and evaluate the effectiveness of R-DXd.

DETAILED DESCRIPTION:
R-DXd is an antibody drug conjugate that specifically binds to CDH6 on the cell surface of target cells, which leads to the internalization of R-DXd into the cells. MAAA-1181a that is released from R-DXd in the target cells inhibits cell replication and induces cell apoptosis.

This study will evaluate R-DXd given as a single agent once every 21 days. The dose escalation phase will enroll participants with OVC and RCC, and is designed to assess the safety and tolerability of R-DXd and to determine the maximum tolerated dose (MTD)/recommended dose for expansion (RDE). Following the selection of the RDE, the dose expansion phase will be initiated to evaluate clinical activity of R-DXd.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* At least 18 years of age
* Eastern Cooperative Oncology Group Performance Status score of 0 or 1
* Availability of archived tumor tissue samples
* Has a left ventricular ejection fraction (LVEF) ≥50% by either an echocardiogram (ECHO) or multigated acquisition scan (MUGA) within 28 days before start of study treatment
* Has adequate organ function within 7 days before the start of study treatment
* Has an adequate treatment washout period prior to start of study treatment
* Male participants with female partners of childbearing potential and female participants of child-bearing potential must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 4 months (for males) and for at least 7 months (for females) after the last dose of study drug.

Exclusion Criteria:

* Has had prior treatment with other CDH6-targeted agents
* Has had prior treatment with an ADC that consists of an exatecan derivative that is a topoisomerase I inhibitor (e.g., trastuzumab deruxtecan, datopotamab deruxtecan, ifinatamab deruxtecan, DS-3939)
* Has history or current presence of CNS metastases except for participants who have completed radiotherapy or surgery ≥2 weeks before the start of study treatment and have no evidence of disease progression in the CNS and no requirement for chronic corticosteroid therapy within 2 weeks before the start of study treatment
* Has multiple primary malignancies, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated, with no evidence of disease for ≥3 years)
* Has a history of myocardial infarction or unstable angina within 6 months before start of study treatment
* Has a medical history of symptomatic congestive heart failure (New York Heart Association classes II-IV) or a cardiac arrhythmia requiring treatment
* Lung-specific intercurrent clinically significant illnesses
* Has an uncontrolled infection requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting toxicities (DLTs) | Day 1 to Day 21 in Cycle 1 (each cycle is 21 days)
Number of Participants Reporting Treatment-emergent Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest | From start of treatment up to 40 days after last dose, up to approximately 52 months
Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) (Dose Expansion) | From start of treatment (Cycle 1, Day 1) up to disease progression, up to approximately 52 months (each cycle is 21 days)
  ORR is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Pharmacokinetic Analysis Area Under the Plasma Concentration-Time Curve from Time Zero to 21 Days (AUC 21d) for R-DXd and its Metabolites | Cycles 1 and 3, Day 1: Predose, 3 hours, 5 hours, 8 hours postdose, end of infusion (EOI); Cycles 1 and 3, Day 2; Cycles 1 and 3, Days 4, 8, and 15; Cycle 2, Day 1: predose and EOI; Cycle 4, Day 1 and every then 2 cycles: predose (each cycle is 21 days)
Pharmacokinetic Analysis Area Under the Plasma Concentration-Time Curve Up to the Last Quantifiable Time (AUClast) for R-DXd and its Metabolites | Cycles 1 and 3, Day 1: Predose, 3 hours, 5 hours, 8 hours postdose, end of infusion (EOI); Cycles 1 and 3, Day 2; Cycles 1 and 3, Days 4, 8, and 15; Cycle 2, Day 1: predose and EOI; Cycle 4, Day 1 and every then 2 cycles: predose (each cycle is 21 days)
Pharmacokinetic Analysis Maximum Plasma Concentration (Cmax) for R-DXd and its Metabolites | Cycles 1 and 3, Day 1: Predose, 3 hours, 5 hours, 8 hours postdose, end of infusion (EOI); Cycles 1 and 3, Day 2; Cycles 1 and 3, Days 4, 8, and 15; Cycle 2, Day 1: predose and EOI; Cycle 4, Day 1 and then every 2 cycles: predose (each cycle is 21 days)
Pharmacokinetic Analysis Lowest Plasma Concentration (Ctrough) for R-DXd and its Metabolites | Cycles 1 and 3, Day 1: Predose, 3 hours, 5 hours, 8 hours postdose, end of infusion (EOI); Cycles 1 and 3, Day 2; Cycles 1 and 3, Days 4, 8, and 15; Cycle 2, Day 1: predose and EOI; Cycle 4, Day 1 and then every 2 cycles: predose (each cycle is 21 days)
Pharmacokinetic Analysis Time to Maximum Plasma Concentration (Tmax) for R-DXd and its Metabolites | Cycles 1 and 3, Day 1: Predose, 3 hours, 5 hours, 8 hours postdose, end of infusion (EOI); Cycles 1 and 3, Day 2; Cycles 1 and 3, Days 4, 8, and 15; Cycle 2, Day 1: predose and EOI; Cycle 4, Day 1 and then every 2 cycles: predose (each cycle is 21 days)
Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Per Investigator and Blinded Independent Central Review (Dose Escalation) | From start of treatment (Cycle 1, Day 1) up to disease progression, up to approximately 52 months (each cycle is 21 days)
  ORR is defined as the proportion of participants with best overall response (BOR) of complete response (CR) or partial response (PR).
Duration of Response (DoR) Based on RECIST v1.1 Per Investigator and Blinded Independent Central Review | From date of first documented response to date of progression or death due to any cause (whichever occurs first), up to approximately 52 months
  DoR is defined as the duration from the first documented response to the date of progression or death due to any cause.
Disease Control Rate (DCR) Based on RECIST v1.1 Per Investigator and Blinded Independent Central Review | From start of treatment up to first documented response (CR, PR, or SD), disease progression, or death (due to any cause), up to approximately 52 months
  DCR is defined as the proportion of participants with BOR of CR, PR, or SD.
Clinical Benefit Rate (CBR) Based on RECIST v1.1 Per Investigator and Blinded Independent Central Review | From date of first documented response (CR, PR) whichever occurs first or SD lasting at least 180 days to disease progression or death (due to any cause), up to approximately 52 months
  CBR is defined as the proportion of participants with BOR of CR or PR, or participants with stable disease (SD) lasting at least 180 days.
Time to Response (TTR) Based on RECIST v1.1 Per Investigator and Blinded Independent Central Review | From start of treatment up to first documented response (CR, PR, or SD), disease progression, or death (due to any cause), up to approximately 52 months
Progression-free Survival Based on RECIST v1.1 Per Investigator and Blinded Independent Central Review | From start of treatment up to disease progression or death (due to any cause), up to approximately 52 months
Percentage of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) and Percentage of Participants Who Have Treatment-emergent ADA | Cycle 1 Day 1, Cycle 1 Day 15, and pre-dose on Day 1 of Cycle 2 through Cycle 4; then every 2 cycles from Cycle 4 through the end of treatment visit (each cycle is 21 days), and 40-day safety follow up visit, up to approximately 52 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (13):
- United States (6):
  - Arizona Oncology Associates, PC HOPE (A)A HOPE), Tucson, Arizona
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Florida Cancer Lake Mary, Lake Mary, Florida
  - Oklahoma University, Oklahoma City, Oklahoma
  - SCRI Oncology Partners, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Japan (7):
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - National Cancer Center Hospital East, Kashiwa-shi, Tokyo
  - National Hospital Organization Kyusyu Cancer Center, Fukuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Kōtoku
  - National Hospital Organization Shikoku Cancer Center, Matsuyama
  - Shizuoka Cancer Center, Nakatogari
  - Saitama Medical University International Medical Center, Saitama

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/